CLINICAL TRIAL: NCT05651620
Title: Legacy Effects of CALERIE™, a 2-year Calorie Restriction Intervention, on Hallmarks of Healthspan and Aging
Brief Title: The CALERIE™ Legacy Study
Status: Active, not recruiting | Type: Observational
Sponsor: Tufts University (Other)
Collaborators: Pennington Biomedical Research Center (Other); Washington University School of Medicine (Other); Duke University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Sai Krupa Das, Professor, Tufts University
Other Study IDs: STUDY00002577; 1R01AG071717-01A1 (NIH)
Record Dates: First submitted 2022-09-01; First posted 2022-12-15 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Calorie Restriction
Keywords: calorie restriction; dietary intervention; biological aging; behavioral data

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood (whole blood, plasma, serum, buffy coat, red blood cells) and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Calorie Restriction (CR): Individuals in the CR group were prescribed a 25% reduction from their baseline energy intake during the two-year CALERIE trial.
- Ad Libitum (AL): Individuals in the AL group were asked to continue their usual dietary intake during the two-year CALERIE trial.

SUMMARY:
The purpose of the CALERIE Legacy Study is to follow up on the health and wellness of participants from phase 2 of the Comprehensive Assessment of Long-term Effects of Reducing Intake of Energy (CALERIE) trial, which was conducted from 2007 to 2011.

DETAILED DESCRIPTION:
The CALERIE Legacy Study is an observational follow-up study of participants from phase 2 the CALERIE trial, the first randomized controlled trial of calorie restriction (CR) in humans without obesity. The overarching goal of the CALERIE Legacy Study is to examine whether two years of CR results in sustained improvements in the biological, phenotypic, and functional hallmarks of human aging 10 to 15 years after the structured intervention. Participants will complete clinical assessments, dietary recalls, and questionnaires, and laboratory evaluations will be performed on blood and urine samples. The study also includes an optional biospecimen banking component.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the CALERIE trial and started their allocated group (CR intervention or ad libitum control condition)
* Willing and able to attend one of the clinical sites for an in-person visit and provide informed consent

Exclusion Criteria:

* Pregnant women
* Women less than 12 months postpartum
* Documented note from the CALERIE trial indicating that the subject should not be contacted or requested not to be contacted for future research
* Diagnosed active cancer or terminal illness

Ages: 33 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All CALERIE participants, except those who are deceased, are known not to qualify, or did not start their allocated group (CR intervention or ad libitum control) (n = 4), have been identified as potential subjects (n = 216) in the CALERIE Legacy Study. The demographic profile of this study is expected to be similar to that of the CALERIE trial, which was 70.4% female. Healthy individuals without obesity of either sex and all race and ethnic groups were eligible to participate in the CALERIE trial. However, due to safety concerns, pregnant women were excluded, and to avoid confounding from peri- and post-menopausal status, the upper age limit for women was 47 years. Upon enrollment, CALERIE participants were 21-50y, 77.3% White, 12% Black, and 10.7% other; ethnicity was 97% non-Hispanic.
Sampling Method: Non-Probability Sample
Enrollment: 216 (Estimated)
Dates: Start 2023-04-06 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Biological age - Klemera-Doubal Method | 10-15 years post CALERIE trial
  Biological age will be quantified by the Klemera-Doubal Method (KDM), an algorithm-based measure. Biological age is expressed in years.
Healthspan | 10-15 years post CALERIE trial
  Healthspan will be assessed by sex-specific metabolic syndrome score (MSS). MSS was developed using mean blood pressure (MBP; = [2 × diastolic blood pressure + systolic blood pressure]/3), high density lipoprotein cholesterol (HDL), triglycerides (TG), waist circumference (WC), and fasting blood glucose (FBG):
  Women: MSS = [45-HDL]/SDHDLW+ [TG-150]/SDTG + [WC-88]/SDWCW + [FBG-100]/SDFBG + [mean BP-100]/SDMBP
  Men: MSS = [40-HDL]/SDHDLW+ [TG-150]/SDTG + [WC-102]/SDWCW + [FBG-100]/SDFBG + [mean BP-100]/SDMBP
  This score does not have a unit.

SECONDARY OUTCOMES:
Height | 10-15 years post CALERIE trial
  Height will be measured in cm.
Weight | 10-15 years post CALERIE trial
  Weight will be measured in kg.
Waist circumference | 10-15 years post CALERIE trial
  Weight circumference will be measured in cm.
Hip circumference | 10-15 years post CALERIE trial
  Hip circumference will be measured in cm.
Body mass index (BMI) | 10-15 years post CALERIE trial
  BMI (kg/m2) will be calculated using height and weight measurements.
Blood pressure | 10-15 years post CALERIE trial
  Systolic and diastolic blood pressure will be measured in mmHg.
Pulse rate at rest | 10-15 years post CALERIE trial
  Pulse rate will be measured in beats/min.
Respiration rate at rest | 10-15 years post CALERIE trial
  Respiration rate will be measured in breaths/min.
Fat mass | 10-15 years post CALERIE trial
  Whole-body fat mass (%) as measured by dual-energy X-ray absorptiometry.
Fat-free mass | 10-15 years post CALERIE trial
  Whole-body fat-free mass (%) as measured by dual-energy X-ray absorptiometry.
Bone mineral content | 10-15 years post CALERIE trial
  Whole-body bone mineral content (g/cm2) as measured by dual-energy X-ray absorptiometry.
Resting metabolic rate (RMR) | 10-15 years post CALERIE trial
  RMR will be measured in kcal/d by indirect calorimetry using a ventilated hood system.
Respiratory quotient (RQ) | 10-15 years post CALERIE trial
  RQ will be measured by indirect calorimetry using a ventilated hood system. This is a ratio and does not have a unit.
Maximal aerobic capacity (V̇O2max) | 10-15 years post CALERIE trial
  Maximal aerobic capacity (V̇O2max) will be measured in mL/kg/min using the Cornell incremental treadmill test.
Interleukin-6 (IL-6) | 10-15 years post CALERIE trial
  IL-6, a blood-based biomarker of aging proposed by the Targeting Aging with MEtformin (TAME) Biomarkers Workgroup, will be measured in pg/mL.
Insulin - TAME panel | 10-15 years post CALERIE trial
  Insulin, a blood-based biomarker of aging proposed by the TAME Biomarkers Workgroup, will be measured in μIU/mL.
Insulin - 0 min (OGTT) | 10-15 years post CALERIE trial
  Insulin (μIU/mL) will be measured at 0 minutes (pre-dose) during an oral glucose tolerance test (OGTT) to evaluate glucoregulatory response.
Insulin - 30 min (OGTT) | 10-15 years post CALERIE trial
  Insulin (μIU/mL) will be measured at 30 minutes post dose during an OGTT to evaluate glucoregulatory response.
Insulin - 60 min (OGTT) | 10-15 years post CALERIE trial
  Insulin (μIU/mL) will be measured at 60 minutes post dose during an OGTT to evaluate glucoregulatory response.
Insulin - 90 min (OGTT) | 10-15 years post CALERIE trial
  Insulin (μIU/mL) will be measured at 90 minutes post dose during an OGTT to evaluate glucoregulatory response.
Insulin - 120 min (OGTT) | 10-15 years post CALERIE trial
  Insulin (μIU/mL) will be measured at 120 minutes post dose during an OGTT to evaluate glucoregulatory response.
Insulin-like growth factor 1 (IGF-1) | 10-15 years post CALERIE trial
  IGF-1, a blood-based biomarker of aging proposed by the TAME Biomarkers Workgroup, will be measured in ng/mL.
Hemoglobin A1c (HbA1c) | 10-15 years post CALERIE trial
  HbA1c, a blood-based biomarker of aging proposed by the TAME Biomarkers Workgroup, will be measured in mmol/mol.
Tumor necrosis factor α receptor II (TNFRII) | 10-15 years post CALERIE trial
  TNFRII, a blood-based biomarker of aging proposed by the TAME Biomarkers Workgroup, will be measured in ng/mL.
High-sensitivity C-reactive protein (hsCRP) | 10-15 years post CALERIE trial
  hsCRP, a blood-based biomarker of inflammation, will be measured in μg/mL.
Growth/differentiation factor 15 (GDF15) | 10-15 years post CALERIE trial
  GDF15, a blood-based biomarker of aging proposed by the TAME Biomarkers Workgroup, will be measured in pg/mL.
Cystatin C | 10-15 years post CALERIE trial
  Cystatin C, a blood-based biomarker of aging proposed by the TAME Biomarkers Workgroup, will be measured in mg/L.
N-terminal B-type natriuretic peptide (NT-proBNP) | 10-15 years post CALERIE trial
  NT-proBNP, a blood-based biomarker of aging proposed by the TAME Biomarkers Workgroup, will be measured in pg/mL.
Senescence-associated secretory phenotype (SASP) proteins | 10-15 years post CALERIE trial
  SASP proteins, blood-based biomarkers of cellular senescence, will be measured using a SASP panel.
Urinary Isoprostanes - iPF(2α)-III | 10-15 years post CALERIE trial
  Urinary iPF(2α)-III, a biomarker of systemic oxidative stress, will be measured in ng/mL.
Urinary Isoprostanes - 2,3-dinor-iPF(2α)-III | 10-15 years post CALERIE trial
  Urinary 2,3-dinor-iPF(2α)-III, a biomarker of systemic oxidative stress, will be measured in ng/mL.
Urinary Isoprostanes - iPF(2α)-VI | 10-15 years post CALERIE trial
  Urinary iPF(2α)-VI, a biomarker of systemic oxidative stress, will be measured in ng/mL.
Urinary Isoprostanes - 8,12-iso-iPF(2α)-VI | 10-15 years post CALERIE trial
  Urinary 8,12-iso-iPF(2α)-VI, a biomarker of systemic oxidative stress, will be measured in ng/mL.
Creatinine | 10-15 years post CALERIE trial
  Creatinine, a byproduct of routine activity in the muscle, will be measured in urine in mg/mL.
Dehydroepiandrosterone (DHEA) | 10-15 years post CALERIE trial
  DHEA, a blood-based steroid hormone, will be measured in μg/dL.
Interleukin 1 beta (IL-1b) | 10-15 years post CALERIE trial
  IL-1b, a blood-based marker of inflammation, will be measured in pg/mL.
Interleukin 8 (IL-8) | 10-15 years post CALERIE trial
  IL-8, a blood-based marker of inflammation, will be measured in pg/mL.
Tumor necrosis factor α (TNF-α) | 10-15 years post CALERIE trial
  TNF-α, a blood-based marker of inflammation, will be measured in pg/mL.
Insulin-like growth factor-binding protein 1 (IGFBP-1) | 10-15 years post CALERIE trial
  IGFBP-1, a blood-based transport protein, will be measured in ng/mL.
Transforming growth factor beta 1 (TGFB1) | 10-15 years post CALERIE trial
  TGFB1, a blood-based marker of immune function, will be measured in ng/mL.
Insulin-like growth factor-binding protein 3 (IGFBP-3) | 10-15 years post CALERIE trial
  IGFBP-3, a blood-based transport protein, will be measured in ng/mL.
Platelet-derived growth factor-AB (PDGF-AB) | 10-15 years post CALERIE trial
  PDGF-AB, a blood-based marker of cellular function, will be measured in ng/mL.
Intercellular Adhesion Molecule 1 (ICAM-1) | 10-15 years post CALERIE trial
  ICAM-1, a blood-based marker of inflammation, will be measured in ng/mL.
Growth hormone | 10-15 years post CALERIE trial
  Growth hormone, a blood-based bio-marker of cellular function, will be measured in ng/mL.
Monocyte Chemoattractant Protein 1 (MCP1) | 10-15 years post CALERIE trial
  MCP1, a blood-based marker of inflammation, will be measured in pg/mL.
Leptin | 10-15 years post CALERIE trial
  Leptin, a hormonal regulator of energy balance, will be measured in pg/mL.
Total adiponectin | 10-15 years post CALERIE trial
  Total adiponectin, a protein hormone that regulates several metabolic processes, including glucose regulation and fatty acid oxidation, will be measured in μg/mL.
High molecular weight adiponectin | 10-15 years post CALERIE trial
  High molecular weight adiponectin, a protein hormone that regulates several metabolic processes, including glucose regulation and fatty acid oxidation, will be measured in μg/mL.
Muscle strength - Knee extension (60°) | 10-15 years post CALERIE trial
  Knee extension at 60 degrees per second will be expressed in Nm.
Muscle strength - Knee extension (180°) | 10-15 years post CALERIE trial
  Knee extension at 180 degrees per second will be expressed in Nm.
Muscle strength - Knee flexion (60°) | 10-15 years post CALERIE trial
  Knee flexion at 60 degrees per second will be expressed in Nm.
Muscle strength - Knee flexion (180°) | 10-15 years post CALERIE trial
  Knee flexion at 180 degrees per second will be expressed in Nm.
Handgrip Strength | 10-15 years post CALERIE trial
  Handgrip strength will be measured via a hand dynamometer and expressed in kg.
Physical functioning | 10-15 years post CALERIE trial
  Physical functioning as measured by a physical performance battery. This physical performance battery provides a composite score ranging from 0 to 12 and includes results from the balance, gait and chair stand tests.
Cognition | 10-15 years post CALERIE trial
  Cognition as measured by the Cambridge Neuropsychological Test Automated Battery (CANTAB). The CANTAB evaluates six main areas of cognitive function: reaction time; verbal recognition memory; intra-extra dimensional set shift; rapid visual information processing; delayed matching to sample; and spatial working memory.
Dietary intake- calories | 10-15 years post CALERIE trial
  Dietary intake in calories (kcals/day), as measured by multiple-pass 24-hour dietary recalls and Nutrition Data System for Research (NDSR) software.
Dietary intake - carbohydrates | 10-15 years post CALERIE trial
  Dietary carbohydrate as % of energy or grams will be measured by multiple-pass 24-hour dietary recalls and Nutrition Data System for Research (NDSR) software.
Dietary intake - proteins | 10-15 years post CALERIE trial
  Dietary proteins as % of energy or grams will be measured by multiple-pass 24-hour dietary recalls and Nutrition Data System for Research (NDSR) software.
Health-related quality of life | 10-15 years post CALERIE trial
  Quality of life as measured by the RAND 36-Item Short Form Survey (SF-36). The RAND SF-36 measures eight aspects of health: physical functioning, role limitations due to physical health problems, role limitations due to personal or emotional problems, energy/fatigue, emotional well-being, social functioning, bodily pain, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. Each item is on a 3- or 5-point Likert scale (1-3 or 1-5). Each response is transformed to a recoded value of 0-100, and the transformed scores of the 9 subscales are averaged to derive a composite score. Higher scores indicate more favorable health states.
Depression status | 10-15 years post CALERIE trial
  Depression status as measured by the Beck Depression Inventory II (BDI-II). The 21-item BDI-II measures depression severity. The score range is 0-63, with higher scores indicating greater depression severity. Nineteen items are on a 4-point Likert scale (0-3). Two items are on a 7-point Likert scale, and responses are scaled to 0-3. The values are summed to calculate the total score.
Mood | 10-15 years post CALERIE trial
  Mood as measured by the Profile of Mood States Second Edition (POMS 2). The POMS 2 assesses six mood subscales using 65 items, each on a 5-point Likert scale (0-4): tension-anxiety (9 items, score range 0-36), depression-dejection (15 items, range 0-60), anger-hostility (12 items, range 0-48), vigor-activity (8 items, range 0-32), fatigue-inertia (7 items, range 0-28), and confusion-bewilderment (7 items, range 0-28). High vigor-activity scores reflect a good mood or emotion, and low scores in the other subscales reflect a good mood or emotion. Total mood disturbance, which is calculated by subtracting the vigor subscale score from the total subscale score (range 0-200), also will be assessed.
Sleep | 10-15 years post CALERIE trial
  Sleep as measured by the Pittsburgh Sleep Quality Index (PSQI). The PSQI measures sleep quality and disturbance over the course of one month using seven subscales: subjective sleep quality; sleep latency; sleep duration; habitual sleep efficiency; sleep disturbances; use of sleeping medication; and daytime dysfunction. The scoring range of each subscale is 0-3. The scoring range of the Global PSQI (the composite score of the seven subscales) is 0-21. For both the subscales and Global PSQI, higher scores indicate greater difficulties with sleeping.
Sexual function | 10-15 years post CALERIE trial
  Sexual function as measured by the Derogatis Interview for Sexual Functioning - Self Report (DISF-SR). Both versions of the DISF-SR (male and female) are scored from 20 to 75, with higher scores indicating higher sexual functioning.
Food cravings | 10-15 years post CALERIE trial
  Food cravings as measured by the Food Cravings Questionnaire-Trait (FCQ-T). The FCQ-T measures frequency and intensity of food cravings. It has 39 items on a 6-point Likert scale (1-6) and a score range of 39-234. Higher scores indicate more frequent and intense food cravings. Scores on all items are summed for a total score.
Dietary restraint, disinhibition, and hunger | 10-15 years post CALERIE trial
  Dietary restraint, disinhibition, and hunger as measured by the Three-Factor Eating Questionnaire (TFEQ). The 51-item TFEQ will be used to measure dietary restraint (21 items), disinhibition (16 items), and hunger (14 items). Item responses are scored as 0 or 1 and summed. Higher scores indicate higher levels of restrained eating (range 0-21), disinhibited eating (range 0-16), and predisposition to hunger (range 0-14).
Disordered eating | 10-15 years post CALERIE trial
  Disordered eating as measured by the Multiaxial Assessment of Eating Disorder Symptoms (MAEDS). MAEDS will be used to assess six domains of disordered eating: binge eating (range 8-56), restrictive eating (range 9-63), purgative behavior (range 7-49), fear of fatness (range 11-77), avoidance of forbidden foods (range 10-70), and depression (range 11-77).
Body shape perceptions | 10-15 years post CALERIE trial
  Body shapes perceptions as measured by the Body Shape Questionnaire (BSQ). Items on the BSQ are rated on a 6-point Likert-type scale. The score ranges from 34-204 points. Higher scores indicate increased concern regarding body shape.
Physical activity | 10-15 years post CALERIE trial
  Physical activity as measured by the 7-Day Stanford Physical Activity Recall (PAR). The PAR estimates an individual's time spent in sleep and physical activity for the 7 days prior to the interview. Energy expenditure based on time spent in sleep and physical activities can be estimated. Sub-scores of energy expenditure for each of the following activities are calculated, summed, and averaged to estimate energy expenditure as kilocalories per day: sleep, moderate physical activity, hard physical activity, and very hard physical activity. Higher scores indicate greater physical activity per day. Metabolic equivalent (MET) value for each activity is provided: 1 MET for sleep, 4 METs for moderate activity, 6 METs for hard activity, and 10 METs for very hard activity. Time spent in each activity over 7 days is multiplied by the appropriate MET value. The minimum value for each activity is zero; there is no maximum value.
Resilience | 10-15 years post CALERIE trial
  Resilience as measured by the 25-item Connor-Davidson Resilience Scale (CD-RISC-25). CD-RISC-25 is scored from 0 to 100, with higher scores indicating higher resilience.
Total cholesterol | 10-15 years post CALERIE trial
  Total cholesterol will be measured in mg/dL using a standard lipid panel.
High-density lipoprotein cholesterol (HDL-C) | 10-15 years post CALERIE trial
  HDL-C will be measured in mg/dL using a standard lipid panel.
Triglycerides | 10-15 years post CALERIE trial
  Triglycerides will be measured in mg/dL using a standard lipid panel.
Low-density lipoprotein cholesterol (LDL-C) | 10-15 years post CALERIE trial
  LDL-C will be calculated in mg/dL using measured values of total cholesterol, HDL-C, and triglycerides.
Glucose - 0 min (OGTT) | 10-15 years post CALERIE trial
  Glucose (mg/dL) will be measured at 0 minutes (pre-dose) during an OGTT to evaluate glucoregulatory response.
Glucose - 30 min (OGTT) | 10-15 years post CALERIE trial
  Glucose (mg/dL) will be measured at 30 minutes post dose during an OGTT to evaluate glucoregulatory response.
Glucose - 60 min (OGTT) | 10-15 years post CALERIE trial
  Glucose (mg/dL) will be measured at 60 minutes post dose during an OGTT to evaluate glucoregulatory response.
Glucose - 90 min (OGTT) | 10-15 years post CALERIE trial
  Glucose (mg/dL) will be measured at 90 minutes post dose during an OGTT to evaluate glucoregulatory response.
Glucose - 120 min (OGTT) | 10-15 years post CALERIE trial
  Glucose (mg/dL) will be measured at 120 minutes post dose during an OGTT to evaluate glucoregulatory response.
Insulin resistance | 10-15 years post CALERIE trial
  Insulin resistance will be calculated using the Homeostatic Model Assessment (HOMA) and measured values of fasting glucose (mmol/L) and fasting insulin (μ/L): (fasting glucose × fasting insulin) ∕ 22.5
Beta-cell function | 10-15 years post CALERIE trial
  Beta-cell function will be calculated using HOMA-β and measures of fasting insulin (μ/L) and fasting glucose (mg/dL): HOMA-β (%) = (360 × fasting insulin) ∕ (fasting glucose - 63)
Triiodothyronine (T3) | 10-15 years post CALERIE trial
  T3, a blood-based marker of thyroid function, will be measured in ng/dL.
Thyroxine (T4) | 10-15 years post CALERIE trial
  T4, a blood-based marker of thyroid function, will be measured in ng/dL.
Thyroid stimulating hormone (TSH) | 10-15 years post CALERIE trial
  TSH, a blood-based marker of thyroid function, will be measured in μIU/mL.
Alkaline phosphatase (ALKP) | 10-15 years post CALERIE trial
  ALKP, a blood-based marker of liver function, will be measured in IU/L.
Alanine transaminase (ALT) | 10-15 years post CALERIE trial
  ALT, a blood-based marker of liver function, will be measured in U/L.
Aspartate aminotransferase (AST) | 10-15 years post CALERIE trial
  AST, a blood-based marker of liver function, will be measured in U/L.
Albumin | 10-15 years post CALERIE trial
  Albumin, a blood-based marker of liver and kidney function, will be measured in g/dL.
Blood Urea Nitrogen (BUN) | 10-15 years post CALERIE trial
  BUN, a blood-based marker of kidney function, will be measured in mg/dL.
Total Proteins | 10-15 years post CALERIE trial
  Total proteins is a measurement sum of albumin and globulin. Total proteins is indicative of blood vessel and immune system function. It will be measured in g/dL.
Bilirubin | 10-15 years post CALERIE trial
  Bilirubin, a blood-based marker of liver function, will be measured in mg/dL.
Creatine Phosphokinase (CPK) | 10-15 years post CALERIE trial
  CPK, an enzyme marker of energy homeostasis, will be measured in U/L.
Lactate Dehydrogenase (LDH) | 10-15 years post CALERIE trial
  LDH, an enzyme marker of liver function, will be measured in U/L.
Globulin | 10-15 years post CALERIE trial
  Globulin, a blood-based marker of liver function, will be measured in g/dL.
Albumin/Globulin (A/G) ratio | 10-15 years post CALERIE trial
  A/G ratio is a blood-based marker used to monitor nutritional status and immune system, kidney, and liver function. This marker is a ratio, and therefore does not have units.
Uric Acid | 10-15 years post CALERIE trial
  Uric acid, a blood-based marker of purine metabolism, will be measured in mg/dL.
Calcium (Ca) | 10-15 years post CALERIE trial
  Calcium, a blood-based mineral, will be measured in mg/dL.
Phosphorus (P) | 10-15 years post CALERIE trial
  Phosphorus, a blood-based mineral, will be measured in mg/dL.
Magnesium (Mg) | 10-15 years post CALERIE trial
  Magnesium, a blood-based mineral, will be measured in meq/L.
Sodium (Na+) | 10-15 years post CALERIE trial
  Sodium, an electrolyte that reflects the body's fluid balance, will be measured in meq/L.
Potassium (K+) | 10-15 years post CALERIE trial
  Potassium, an electrolyte that reflects the body's fluid balance, will be measured in meq/L.
Chloride (Cl-) | 10-15 years post CALERIE trial
  Chloride, an electrolyte that reflects the body's fluid balance, will be measured in meq/L.
Apoprotein A1 | 10-15 years post CALERIE trial
  Apoprotein A1, a blood-based marker of lipid metabolism, will be measured in mg/dL.
Apoprotein B | 10-15 years post CALERIE trial
  Apoprotein B, a blood-based marker of lipid metabolism, will be measured in mg/dL.
Biological age - Homeostatic Dysregulation | 10-15 years post CALERIE trial
  Biological age will be quantified by homeostatic dysregulation, an algorithm-based measure. Biological age is expressed in years.
Biological age - Levine Phenotypic Age | 10-15 years post CALERIE trial
  Biological age will be quantified by Levine Phenotypic Age, an algorithm-based measure. Biological age is expressed in years.

CONTACTS AND LOCATIONS:
Overall Officials: Sai Krupa Das, PhD, Principal Investigator — Tufts University
Locations (3):
- United States (3):
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: Yes
Per the NIH Data Public Access Policy, after study closure, the data coordinating center at Duke University will lock the electronic database and clean and deidentify the data prior to public posting. Biospecimens collected for banking will be deidentified and transferred to the NIA AgingResearchBiobank, which utilizes a state-of-the-art inventory system for the storage and distribution of study samples for future scientific research.
  The study protocol and informed consent form will be made available as well.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be posted for open access use at the time of publication of the primary manuscript. Biospecimens will be stored at the NIA Biobank and will be available upon study completion and until all samples are depleted or deemed not viable.
Access Criteria: Permission to use data will not be restricted. However, interested investigators must register with the applicable website to access data, which will be made available via download. Data collected in this study will be appropriate for regression adapted to longitudinal data and multivariate-multivariable analysis or goodness-of-fit chi-square, non-parametric measures of association.
  Investigators interested in accessing biospecimens will need to apply for access by submitting a request via the NIA AgingResearchBiobank website (https://agingresearchbiobank.nia.nih.gov/how-to-make-a-request/). To submit this request, a designated member of the investigative team will be required to register as a user on the AgingResearchBiobank website. Any investigator can submit a request for access to the biospecimens for future research but must be approved by the AgingResearchBiobank to gain access. Biospecimens will be provided as samples that will be shipped to approved investigators.

DOCUMENTS (1):
  • Informed Consent Form (2025-03-06): https://cdn.clinicaltrials.gov/large-docs/20/NCT05651620/ICF_003.pdf